CLINICAL TRIAL: NCT03125954
Title: Changes in Physical Inactivity Secondary to Exercise Therapy in Patients with Knee Osteoarthritis: a Prospective Cohort Study
Brief Title: Changes in Physical Inactivity in Patients with Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Other Study IDs: InactivityOAIII
Record Dates: First submitted 2017-03-21; First posted 2017-04-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2018-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: standardized exercise treatment for knee OA in Denmark (GLAiD) — objective measurement of physical activity before, during af after the GLAiD intervention

SUMMARY:
This is an objective cohort study using objective recording of physical activity (accelerometry) during and after the GLAiD intervention to investigate if a sedentary behavior change by participating in an 6-week physiotherapy-led exercise and education program (GLAiD) occurs. The GLAiD intervention is an education and exercise based intervention aiming at decreasing pain and improving function in patients with knee osteoarthritis.

The primary outcome is change in objective recorded physical activity between baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years
* Diagnosed with knee OA
* Willing and able to complete study visits and procedures
* Owner of a smartphone or tablet
* Eligible for participation in the GLAID treatment
* Speaks, reads and writes Danish language

Exclusion Criteria:

* Any condition, which in the opinion of the Investigator, would put the subject at increased safety risk by participation, or otherwise make the subject unsuitable for this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with knee osteoarthritis refered to the GLAiD program
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Objectively measured physical activity | 6 weeks
  accelerometer recorded physical activity

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score(KOOS) | baseline (day 1) and follow-up (after 6 weeks)
  KOOS questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bartholdy C, Skou ST, Bliddal H, Henriksen M. Changes in physical inactivity during supervised educational and exercise therapy in patients with knee osteoarthritis: A prospective cohort study. Knee. 2020 Dec;27(6):1848-1856. doi: 10.1016/j.knee.2020.09.007. Epub 2020 Nov 13. PMID 33197825